CLINICAL TRIAL: NCT00065819
Title: HIV Symptom Management With African American Mothers
Brief Title: HIV Symptom Management Program for African American Mothers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NR004416 (NIH); RR000466GCRC
Record Dates: First submitted 2003-08-01; First posted 2003-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: HIV; African American; Symptom Management
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: HIV Symptom Education Program

SUMMARY:
African American mothers infected with HIV face unique challenges in management of their disease. The goal of this study was to determine the effectiveness of an HIV self-care and symptom management program designed to help low-income African American mothers with HIV.

DETAILED DESCRIPTION:
Infection with the human immunodeficiency virus (HIV) poses a growing threat to the health of women in childbearing years and occurs disproportionately among lower socioeconomic populations and minority women. Early identification of HIV infection and advances in antiretroviral therapies have begun to prolong the lives of infected individuals. However, women with HIV appear to have more rapid disease progression and shorter survival after diagnosis than men. Evidence is emerging that women are less likely to use health services, are more likely to present at clinical facilities with advanced disease, and are less likely to receive antiretroviral therapy.

To date, little attention has focused on the prevention and management of symptoms experienced by women with HIV before they develop AIDS. The primary aim of this randomized clinical study was determine the efficacy of an HIV self-care and symptom management intervention designed to help low-income African American mothers with HIV. The study was based on the Maternal HIV Self-Care Symptom Management framework, which postulates that helping mothers to cope with their emotional responses to HIV diagnosis and to reframe their understanding of HIV from an immediate life-threatening illness to a chronic disease decreases emotional distress and improves health.

One hundred and nine African American mothers, including 17 grandmothers who were primary caregivers for children, participated in the trial. Women were randomized to either the intervention or the control group. The intervention focused on the mother's responses to her HIV diagnosis and helped her understand, manage, and prevent selected HIV-related symptoms, using her concern about her child(ren) as a motivator. The intervention used a cognitive reframing educational approach based within a therapeutic relationship with an advanced practice nurse. The nurse provided a culturally sensitive milieu designed to help the woman feel safe in exploring her feelings and expressing her needs. Eight teaching modules provided basic information to improve knowledge about HIV and help the mother identify self-care strategies related to general health promotion. Data were collected using self-report measures assessing emotional distress and health.

Mothers in the intervention group reported fewer feelings of stigma 6 months after the intervention ended than did mothers in the control group. Within the intervention group, there was a reduction in two aspects of affective state (depression/dejection and tension/anxiety) and in stigma. However, most outcomes did not differ significantly. There was no reduction in depressive symptoms, in other aspects of affective state, or in HIV worry. Mothers in the intervention group reported higher physical function scores 6 months after the intervention ended compared to control mothers. Other aspects of health-related quality of life, such as perception of health, health distress, energy/fatigue, and role function, did not improve. Within the intervention group, mothers reported fewer infections from enrollment to 1 month after the intervention ended. In contrast, mothers in the control group reported a decline in physical function and overall role function. There was a high drop-out for mothers in both groups. Analysis of enrollment data comparing the mothers who dropped out and mothers who remained in the study indicated that drop-out mothers had significantly higher scores on emotional distress variables and social conflict and lower perceptions of health, suggesting the need for a more targeted intervention with a stronger focus on mental health.

ELIGIBILITY:
Inclusion Criteria

* African American
* HIV infected
* Primary caregiver of child(ren) under the age of 9

Exclusion Criteria

* Diagnosis of AIDS

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Margaret S. Miles, RN, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Black BP, Miles MS. Calculating the risks and benefits of disclosure in African American women who have HIV. J Obstet Gynecol Neonatal Nurs. 2002 Nov-Dec;31(6):688-97. doi: 10.1177/0884217502239211. PMID 12465865
- [Background] Mallory C, Miles MS, Holditch-Davis D. Reciprocity and retaining African-American women with HIV in research. Appl Nurs Res. 2002 Feb;15(1):35-41. doi: 10.1053/apnr.2002.29529. PMID 11840408
- [Background] Miles MS, Gillespie JV, Holditch-Davis D. Physical and mental health in African American mothers with HIV. J Assoc Nurses AIDS Care. 2001 Jul-Aug;12(4):42-50. doi: 10.1016/S1055-3290(06)60215-X. PMID 11486719